CLINICAL TRIAL: NCT06199986
Title: De-implementation of Low Value Castration for Men With Prostate Cancer - Living Well With Prostate Cancer
Brief Title: DeADT - Living Well With Prostate Cancer
Acronym: DeADT-LW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Sameer D. Saini, Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1656029; R37CA222885 (NIH)
Record Dates: First submitted 2023-12-19; First posted 2024-01-10 (Actual); Results first posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Veterans
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ADT Order Check Attestation (Or) (Experimental): Study staff will place a "Living Well ADT" health factor in the electronic medical record for patients already receiving ADT, and whose clinic visits the study team have confirmed to be targets for ADT de-implementation. Health factors will be entered as eligible clinic visits are identified. This health factor combined with a low PSA level (most recent PSA < 2) will trigger the ADT Order Check Attestation Intervention (Or) when the provider participant places an order for ADT (e.g., Lupron, Eligard, Goserelin, and Zoladex). Provider participants may override the order check by entering text indicating the reason and continue with the ordering process.
  Interventions: Behavioral: ADT Order Check Attestation (Or)
- Provider Script (Sc) (Experimental): Study staff will enter an electronic health record progress note approximately one business day prior to a target low-value ADT clinic visit from a patient already receiving ADT. The note will include scripted talking points for the provider participant to help with discussion and recent PSA levels and can be edited, signed, or deleted by the provider, giving a quick and simple way to document the discussion. The progress note will prompt provider participants to indicate whether a patient prefers to continue or discontinue ADT. The progress note will include links to a patient-facing clinic handout which will be posted on an external website. Provider participants may modify, ignore, or delete the progress note.
  Interventions: Behavioral: Provider Script (Sc)
- Control (No Intervention): The study team will match up to 8 sites (i.e., medical centers) to the 4 randomized sites as contemporary controls where no interventions have been deployed to compare the primary outcome of interruption of low-value ADT injections. Low-value ADT injections, eligible clinic visits, and primary outcomes for a matched 6-month period will be ascertained through chart review and compared to intervention site primary outcomes.

INTERVENTIONS:
Behavioral: ADT Order Check Attestation (Or) — Clinical reminder order check in electronic health record
  Arms: ADT Order Check Attestation (Or)
Behavioral: Provider Script (Sc) — Provider script added to progress note in electronic health record
  Arms: Provider Script (Sc)

SUMMARY:
The goal of this randomized de-implementation trial is to compare two strategies to reduce low-value androgen deprivation therapy (ADT) use for prostate cancer care. The aim of the study is to compare implementation of the two strategies: use of a clinical reminder order check intervention versus a provider script/patient education approach, and their impacts on low-value ADT use after six months. The main goal of both interventions will be to decrease ADT overuse for patients with prostate cancer, but to do this in a way that is acceptable to the clinicians who treat these patients. The interventions will be initiated for providers only across 4 participating facilities. Provider participants will engage with one of the interventions triggered in the electronic health record when their patients are deemed likely to be receiving low-value ADT. Each provider participant receives only one of the interventions. The intervention is triggered for every clinic visit involving a patient deemed to be receiving low-value ADT, so provider participants may receive their assigned intervention multiple times. Researchers will compare provider use of both strategies to determine implementation outcomes and whether one was more effective in reducing low-value ADT use.

DETAILED DESCRIPTION:
Project Background:

Prostate cancer is a leading male cancer. One in three men with prostate cancer is chemically castrated at some point with long-acting injectable drugs (i.e., androgen deprivation therapy or ADT). Although some patients benefit in terms of survival and symptom improvement, chemical castration with ADT is also commonly performed when there are little to no health benefits to patients raising questions of low-value care and overuse. A growing awareness of castration harms (e.g., heart attack, osteoporosis, loss of sexual function) also creates patient safety concerns. Despite this, ADT use in low-value cases, such as for localized prostate cancer treatment and biochemical recurrence in non-metastatic disease persists.

Ineffective and harmful practices such as chemical castration of prostate cancer patients with ADT outside of the evidence base are ideal targets for de-implementation. De-implementation, or stopping low value practices, has the potential to improve patient outcomes and decrease healthcare costs. For example, stopping low-value chemical castration overuse could prevent harm, limit spending, and maintain survival. However, provider preferences regarding de-implementation are not well understood, and possible de-implementation interventions range from blunt formulary restriction policies to shared decision-making. Blunt policy interventions such as formulary restriction of ADT (e.g., pre-authorization, order templates) might seem warranted given patient safety concerns, yet could result in significant provider resistance and work-arounds if introduced poorly. More nuanced, patient-centered interventions such as shared decision-making (e.g., decision aid, talking points) likely involve extra clinical time. Both intervention strategies need tailoring based on provider input for acceptability and feasibility in clinical practice, including piloting prior to trialing. As many medical practices lack evidence and cause harm, robust, behavioral theory-based methods for incorporating provider preferences into de-implementation strategy development will advance both implementation research and practice.

Project Objectives:

This study will compare two different de-implementation strategies that vary in delivery, impact, and expected results for reducing low-value ADT use.

Research Plan/Methods:

Compare two tailored de-implementation strategies to reduce chemical castration as localized prostate cancer treatment and treatment for non-metastatic biochemical recurrence with low PSA levels.

The specific aim is to evaluate the implementation of an ADT order check (Or) versus a provider script (Sc) on decreased low-value ADT use after six months.

The study team will recruit Site Champions (e.g., Urology Chiefs) at each of the participating sites (i.e., medical centers). All clinicians who prescribe ADT at participating sites will be eligible to receive the interventions. Ann Arbor team members will send clinicians an email with an attached Research Information Sheet providing an opportunity to opt out of participation. Opting out means that they will not be asked to participate in surveys or other approaches to measuring provider responses and the interventions will not be triggered for any of their patients or clinic visits.

No other inclusion or exclusion criteria will be applied. No patients will be recruited for this study; however, identifiable data will be collected from national VA CDW, Central Cancer Registry, and Vital Status data, and chart reviews will be conducted using CPRS/Capri/JLV/ WebVRAM, to identify target clinic visits and assess outcomes. Identifiers will be stripped as early as possible, once analytic data sets are created.

Implementation outcomes will be collected from VA CDW/Cancer Registry/Vital Status records and CPRS/Capri/JLV/WebVRAM for all clinic visits documented as providing low-value ADT at 6 months. An anonymous clinic assessment survey will be administered to Site Champions at baseline and an ADT provider assessment will be administered to participating site providers at baseline and 1-month post-intervention through VA Qualtrics.

Outcomes Analyses

Primary analyses: Comparing the effectiveness of two de-implementation strategies, Or and Sc, on low-value ADT use after six months. The primary outcome is interruption of ADT injections, evaluated through a combination of chart reviews and informatics data generated through the ordering process. The intervention sites were matched with 4 control sites acting as contemporary controls for ADT overuse and effectiveness outcomes.

Secondary outcomes: The secondary outcomes focus on implementation of the strategies and interventions across sites including reach, penetration, and feasibility at site and clinic levels.

ELIGIBILITY:
Inclusion Criteria:

* Any provider at participating sites who prescribes ADT for prostate cancer patients

Exclusion Criteria:

* Providers opting out of study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-10-04 (Actual); Primary Completion 2024-04-16 (Actual); Study Completion 2024-04-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sameer D Saini, MD, Principal Investigator — VA Ann Arbor Healthcare System/University of Michigan
Locations (1):
- VA Ann Arbor Healthcare System, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Members of the scientific community who would like a copy of the de-identified final data sets (i.e., data sets underlying any publication) from this study can request a copy by e-mailing Jennifer Burns at jennifer.burns@va.gov. They should state their reason for requesting the data and their plans for analyzing the data. Final data sets will be copied onto an encrypted CD. The CD will be sent to the requestor via FedEx.
Time Frame: Data will be available once RCT is complete and up to 6 years after the end of the fiscal year in which the project is terminated.
Access Criteria: Members of the scientific community who would like a copy of the de-identified final data sets (i.e., data sets underlying any publication) from this study can request a copy by e-mailing Jennifer Burns at jennifer.burns@va.gov. They should state their reason for requesting the data and their plans for analyzing the data. Final data sets will be copied onto an encrypted CD. The CD will be sent to the requestor via FedEx.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were providers who received the study interventions and are represented by the ADT Order Check Attestation (Or) and Provider Script (Sc) arms.
  Patients were not participants, as they received no interventions, although their data was collected to assess the effect of the interventions on the provider participants. Patients are represented by the ADT Order Check Attestation (Or) - Patients, Provider Script (Sc) - Patients, and Control arms.
Units Other Than Participants: Centers
Groups:
- ADT Order Check Attestation (Or) - Providers; ADT Order Check Attestation (Or) - Patients: Study staff placed a "Living Well ADT" health factor in the electronic medical record for patients already receiving ADT, and whose clinic visits the study team confirmed to be targets for ADT de-implementation. Health factors were entered as eligible clinic visits were identified. This health factor combined with a low PSA level (most recent PSA < 2) triggered the ADT Order Check Attestation Intervention (Or) when the provider participant placed an order for ADT (e.g., Lupron, Eligard, Goserelin, and Zoladex). Provider participants could override the order check by entering text indicating the reason and continue with the ordering process.
  ADT Order Check Attestation (Or): Clinical reminder order check in electronic health record.
- Provider Script (Sc) - Providers; Provider Script (Sc) - Patients: Study staff entered an electronic health record progress note approximately one business day prior to a target low-value ADT clinic visit from a patient already receiving ADT. The note included scripted talking points for the provider participant to help with discussion and recent PSA levels and could be edited, signed, or deleted by the provider, giving a quick and simple way to document the discussion. The progress note prompted provider participants to indicate whether a patient preferred to continue or discontinue ADT. The progress note included links to a patient-facing clinic handout which was posted on an external website. Provider participants could modify, ignore, or delete the progress note.
  Provider Script (Sc): Provider script added to progress note in electronic health record.
- Control: The study team matched 4 sites (i.e., medical centers) to the 4 randomized sites as contemporary controls where no interventions were deployed to compare the primary outcome of interruption of low-value ADT injections. Low-value ADT injections, eligible clinic visits, and primary outcomes for a matched 6-month period were ascertained through chart review and compared to intervention site primary outcomes.
Period: Overall Study
Arm/Group | ADT Order Check Attestation (Or) - Providers | ADT Order Check Attestation (Or) - Patients | Provider Script (Sc) - Providers | Provider Script (Sc) - Patients | Control
Started (Started (in the Clinician Participant "arms") means the number of clinicians who were prescribing ADT prior to the start of the study, and who received an information and opt-out email.) | 36; 2 Centers | 105; 2 Centers | 14; 2 Centers | 99; 2 Centers | 282; 4 Centers
Completed (Completed here is synonymous with Started and was used to calculate the secondary outcome measure: Reach. There is no "subsequent" measure of Completed.) | 36; 2 Centers | 105; 2 Centers | 14; 2 Centers | 99; 2 Centers | 282; 4 Centers
Not Completed | 0; 0 Centers | 0; 0 Centers | 0; 0 Centers | 0; 0 Centers | 0; 0 Centers

BASELINE CHARACTERISTICS:
Population: Baseline data was not collected from any provider participant, i.e., participants in the ADT Order Check Attestation (Or) - Providers arm or the Provider Script (Sc) - Providers arm. Baseline data is provided for patients because some outcome measures relate to their care.
Groups:
- Total: Total of all reporting groups
Arm/Group | ADT Order Check Attestation (Or) - Patients | Provider Script (Sc) - Patients | Control | Total
Number analyzed (Participants) | 105 | 99 | 282 | 486
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Population: Age data was not collected from any provider participant, i.e., participants in the ADT Order Check Attestation (Or), Provider Script (Sc), and Control arms.
  years | 79 [76 to 85] | 76 [72 to 80] | 76 [72.5 to 79.5] | 77 [73.1 to 80.9]
Sex/Gender, Customized [Count of Participants; unit: Participants] — Sex/Gender data was not collected from any provider participant, i.e., participants in the ADT Order Check Attestation (Or), Provider Script (Sc), and Control arms. All patients in the patient arms (ADT Order Check Attestation (Or) - Patient and Provider Script (Sc) - Patient) were male.
  Participants
    Male | 105 | 99 | 282 | 486
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Ethnicity data was not collected from any provider participant, i.e., participants in the ADT Order Check Attestation (Or), Provider Script (Sc), and Control arms.
  Participants
    Hispanic or Latino | 1 | 5 | 26 | 32
    Not Hispanic or Latino | 101 | 89 | 235 | 425
    Unknown or Not Reported | 3 | 5 | 21 | 29
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race data was not collected from any provider participant, i.e., participants in the ADT Order Check Attestation (Or), Provider Script (Sc), and Control arms.
  Participants
    American Indian or Alaska Native | 1 | 0 | 1 | 2
    Asian | 0 | 0 | 2 | 2
    Native Hawaiian or Other Pacific Islander | 2 | 2 | 5 | 9
    Black or African American | 7 | 43 | 92 | 142
    White | 94 | 46 | 156 | 296
    More than one race | 1 | 1 | 2 | 4
    Unknown or Not Reported | 0 | 7 | 24 | 31
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 105 | 99 | 282 | 486

OUTCOME MEASURES:

1. Primary Outcome: Effectiveness - Interruption in Low Value ADT Injection (i.e., Take a Break From ADT)
Description: The proportion of patients receiving ADT whose prescribed ADT injections were interrupted, as shown by count of patients whose injections were interrupted.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | ADT Order Check Attestation (Or) - Patients | Provider Script (Sc) - Patients | Control
Number analyzed (Participants) | 105 | 99 | 282
Participants | 12 | 28 | 24

2. Secondary Outcome: Reach
Description: The percentage of provider participants who have prescribed ADT before, were asked to participate in the study, and did not opt out of the study.
Time Frame: 6 months
Measure: Number; unit: percentage of provider participants
Arm/Group | ADT Order Check Attestation (Or) - Providers | Provider Script (Sc) - Providers
Number analyzed (Participants) | 36 | 14
percentage of provider participants | 100 | 100

3. Secondary Outcome: Penetration - ADT Order Check Attestation (OR) Intervention
Description: Proportion of OR interventions where the provider participant did not override the order check and prescribe ADT. These providers received the education session about the order checks in the study. However, because of technological problems, the order check did not activate within the 6-month study period.
Time Frame: 6 months
Measure: Number; unit: proportion of OR interventions
Units Other Than Participants: Order checks
Arm/Group | ADT Order Check Attestation (Or) - Providers
Number analyzed (Participants) | 36
Number analyzed (Order checks) | 105
proportion of OR interventions | 0

4. Secondary Outcome: Penetration - Provider Script (SC) Intervention
Description: The total number of SC intervention notes assigned to participant providers by the study team that were actually signed by the providers.
Time Frame: 6 months
Population: Of 99 eligible cases, 81 were actually assigned the script progress note because of unavailability of provider visit, missed appointment, or study team not available for note placement.
Measure: Count of Units; unit: notes
Units Other Than Participants: notes
Arm/Group | Provider Script (Sc) - Providers
Number analyzed (Participants) | 14
Number analyzed (notes) | 81
notes | 64

5. Secondary Outcome: Feasibility - Site Level: Medical Center Director (MCD) Approval
Description: The percentage of sites (i.e., medical centers) asked to participate that received MCD approval to implement the intervention (Order Check or Progress Note/Patient Handout). Each site has only one MCD.
Time Frame: Within 1 month of request to participate being sent
Measure: Count of Units; unit: sites
Units Other Than Participants: sites
Arm/Group | ADT Order Check Attestation (Or) - Providers | Provider Script (Sc) - Providers
Number analyzed (Participants) | 36 | 14
Number analyzed (sites) | 2 | 2
sites | 2 | 2

6. Secondary Outcome: Feasibility - Site Level: Fully Operationalized Intervention
Description: The percentage of approved sites with fully operationalized intervention, i.e. intervention programmed into site EHR and ready to be implemented. Depending on randomization arm, this included either health factor placement or script assignment prior to at least one patient visit.
Time Frame: 6 months
Measure: Count of Units; unit: sites
Units Other Than Participants: sites
Arm/Group | ADT Order Check Attestation (Or) - Providers | Provider Script (Sc) - Providers
Number analyzed (Participants) | 36 | 14
Number analyzed (sites) | 2 | 2
sites | 2 | 2

7. Secondary Outcome: Feasibility - Clinic Level Activation: Clinics With Intervention Implementation
Description: The percentage of approved sites with at least 1 intervention implemented, i.e. at least 1 health factor assigned and/or at least 1 progress note assigned to a provider participant.
Time Frame: Within 6 months
Measure: Count of Units; unit: sites
Units Other Than Participants: sites
Arm/Group | ADT Order Check Attestation (Or) - Providers | Provider Script (Sc) - Providers
Number analyzed (Participants) | 36 | 14
Number analyzed (sites) | 2 | 2
sites | 0 | 2

ADVERSE EVENTS:
Time Frame: Clinic participation was approximately six months long but no AE data was collected.
Description: No AE data was collected in any form - as this was just a feasibility study for implementation.
Groups:
- ADT Order Check Attestation (Or); ADT Order Check Attestation (Or) - Patients: Study staff placed a "Living Well ADT" health factor in the electronic medical record for patients already receiving ADT, and whose clinic visits the study team confirmed to be targets for ADT de-implementation. Health factors were entered as eligible clinic visits were identified. This health factor combined with a low PSA level (most recent PSA < 2) triggered the ADT Order Check Attestation Intervention (Or) when the provider participant placed an order for ADT (e.g., Lupron, Eligard, Goserelin, and Zoladex). Provider participants could override the order check by entering text indicating the reason and continue with the ordering process.
  ADT Order Check Attestation (Or): Clinical reminder order check in electronic health record.
- Provider Script (Sc); Provider Script (Sc) - Patients: Study staff entered an electronic health record progress note approximately one business day prior to a target low-value ADT clinic visit from a patient already receiving ADT. The note included scripted talking points for the provider participant to help with discussion and recent PSA levels and could be edited, signed, or deleted by the provider, giving a quick and simple way to document the discussion. The progress note prompted provider participants to indicate whether a patient preferred to continue or discontinue ADT. The progress note included links to a patient-facing clinic handout which was posted on an external website. Provider participants could modify, ignore, or delete the progress note.
  Provider Script (Sc): Provider script added to progress note in electronic health record.
Arm/Group | ADT Order Check Attestation (Or) | ADT Order Check Attestation (Or) - Patients | Provider Script (Sc) | Provider Script (Sc) - Patients | Control
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2023-11-30): https://cdn.clinicaltrials.gov/large-docs/86/NCT06199986/Prot_000.pdf